CLINICAL TRIAL: NCT02314065
Title: Cognitive Behavioral Therapy for Health Anxiety: a Randomized Controlled Non-inferiority Trial of Internet-delivered and Face-to-Face Therapy
Brief Title: Cognitive Behavioral Therapy for Health Anxiety: Internet Treatment Versus Face-to-Face Therapy
Acronym: HA-NonInf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA-NonInf
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Severe Health Anxiety; Somatic Symptom Disorder; Illness Anxiety Disorder
Keywords: Severe health anxiety; Somatic symptom disorder; Illness anxiety disorder; Cognitive behavioral therapy; Internet; Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional CBT (Experimental): Cognitive Behavioural Therapy delivered in a conventional manner
  Interventions: Behavioral: CBT, exposure and response prevention (Face-to-face)
- Internet-delivered CBT (Experimental): Cognitive Behavioural Therapy delivered via the Internet
  Interventions: Behavioral: CBT, exposure and response prevention (Internet-based)

INTERVENTIONS:
Behavioral: CBT, exposure and response prevention (Face-to-face) — This intervention entails different exercises aimed at exposure to health anxiety stimuli.
  Treatment is delivered in a conventional manner. Participants are physically meeting with a therapist once a week.
  Arms: Conventional CBT
Behavioral: CBT, exposure and response prevention (Internet-based) — This intervention entails different exercises aimed at exposure to health anxiety stimuli.
  Treatment is delivered via the Internet. Participants are guided by a therapist using an email-like communication system.
  Arms: Internet-delivered CBT

SUMMARY:
Background

Severe health anxiety is a highly distressing, often debilitating, psychological problem. Since the release of the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) its clinical manifestations are increasingly often referred to as Somatic Symptom Disorder (SSD) or Illness Anxiety Disorder (IAD). Despite often being overlooked in routine care, several treatments for severe health anxiety have shown great promise, the most well-established being Cognitive Behavioral Therapy (CBT). Traditionally, CBT - like most other psychotherapies - has typically been delivered face-to-face. That is, the patient physically meeting with the therapist once a week for the whole of the treatment. Internet-delivered CBT does not rest on this requirement, but has nevertheless been shown to be efficacious for severe health anxiety (see for example NCT01673035).

Aim of the study

The present study aims to compare the effects of Internet-delivered CBT and CBT face-to-face for severe health anxiety in a randomized controlled trial. A non-inferiority criterion is applied to determine if Internet-delivered CBT is at least as efficacious as its well-established predecessor.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of severe health anxiety (somatic symptom disorder or illness anxiety disorder) according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5)
* Registered citizen of Stockholm county
* At least 18 years old

Exclusion Criteria:

* Other primary axis-I disorder
* Substance abuse or addiction during the last 6 months
* Current or previous episode of psychosis or bipolar disorder
* Severe major depressive disorder
* Suicide risk
* Personality disorder making the treatment procedure very difficult
* Non-stable psychiatric pharmacotherapy (dosage changed during the last 2 months) and the drug is likely to affect outcome measures
* Ongoing concurrent psychological treatment for severe health anxiety
* Having received previous high quality Cognitive Therapy or Cognitive Behavioural Therapy during the recent year
* Ongoing serious somatic disorder, precluding CBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Health Anxiety Inventory (HAI) | baseline, post-treatment (12 weeks), weekly during treatment, 6 month follow-up, 12 month follow-up
  Change in HAI at post-treatment and follow-ups compared to baseline. Analyses will be conducted both within an intention-to-treat (ITT) framework and on a complete case basis. A non-inferiority limit of 0.3 d (effect size) will be used.

SECONDARY OUTCOMES:
Illness Attitude Scale (IAS) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in IAS at post-treatment and follow-ups compared to baseline
Whiteley Index (WI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in WI at post-treatment and follow-ups compared to baseline
Montgomery-Åsberg Depression Rating Scale - Self report (MADRS-S) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in MADRS-S at post-treatment and follow-ups compared to baseline
Beck Anxiety Inventory (BAI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in BAI at post-treatment and follow-ups compared to baseline
Anxiety Sensitivity Index (ASI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in ASI at post-treatment and follow-ups compared to baseline
Sheehan Disability Scale (SDS) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in SDS at post-treatment and follow-ups compared to baseline
Trimbos and institute of medical technology assessment cost questionnaire (TIC-P) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in TIC-P at post-treatment and follow-ups compared to baseline
Euroqol-5D (EQ-5D) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in EQ-5D at post-treatment and follow-ups compared to baseline
Insomnia Severity Index (ISI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in ISI at post-treatment and follow-ups compared to baseline
Self-rated health 5 (SRH-5) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in SRH-5 at post-treatment and follow-ups compared to baseline
Quality of Life Inventory (QOLI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in QOLI at post-treatment and follow-ups compared to baseline
Alcohol Use Disorders Identification Test (AUDIT) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in AUDIT at post-treatment and follow-ups compared to baseline
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (12 weeks)
  For assessing satisfaction with treatment
Sickness Questionnaire (SQ) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in SQ at post-treatment and follow-ups compared to baseline
Perceived Vulnerability for Disease (PVD) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in PVD at post-treatment and follow-ups compared to baseline
Disgust Scale-Rev (DS-R) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in DS-R at post-treatment and follow-ups compared to baseline
WHO Disability Assessment Schedule (WHODAS) 2.0, 12-item version | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in WHODAS at post-treatment and follow-ups compared to baseline

OTHER OUTCOMES:
Psychological mediators | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Assessment of whether these mediators will precede change in outcome during the treatment. Mediators will be assessed using sub scales of the Health Anxiety Inventory, the Insomnia Severity Index, Self-Rated Health 5 and Acceptance/Flexibility. Common health anxiety behaviors will also be assessed.
Credibility/Expectancy scale | Weeks 2 and 8
  For assessing treatment credibility and expectancy of improvement
Working Alliance Inventory (WAI) | Weeks 2 and 8
  For assessing therapeutic alliance

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman, Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Gustavsberg primary care clinic, Gustavsberg, Stockholm County, Sweden

REFERENCES:
- [Background] Hedman E, Andersson E, Lindefors N, Andersson G, Ruck C, Ljotsson B. Cost-effectiveness and long-term effectiveness of internet-based cognitive behaviour therapy for severe health anxiety. Psychol Med. 2013 Feb;43(2):363-74. doi: 10.1017/S0033291712001079. Epub 2012 May 21. PMID 22608115
- [Background] Hedman E, Axelsson E, Gorling A, Ritzman C, Ronnheden M, El Alaoui S, Andersson E, Lekander M, Ljotsson B. Internet-delivered exposure-based cognitive-behavioural therapy and behavioural stress management for severe health anxiety: randomised controlled trial. Br J Psychiatry. 2014 Oct;205(4):307-14. doi: 10.1192/bjp.bp.113.140913. Epub 2014 Aug 7. PMID 25104835
- [Background] Olatunji BO, Kauffman BY, Meltzer S, Davis ML, Smits JA, Powers MB. Cognitive-behavioral therapy for hypochondriasis/health anxiety: a meta-analysis of treatment outcome and moderators. Behav Res Ther. 2014 Jul;58:65-74. doi: 10.1016/j.brat.2014.05.002. Epub 2014 May 24. PMID 24954212
- [Background] Furer P, Walker JR. Treatment of Hypochondriasis with Exposure. Journal of Contemporary Psychotherapy 35(3): 251-267, 2005.
- [Derived] Axelsson E, Osterman S, Hedman-Lagerlof E. Joint factor analysis and approximate equipercentile linking of common trait health anxiety measures: a cross-sectional study of the 14-, 18- and 64-item health anxiety inventory, the illness attitude scale, and the 14-item Whiteley Index. BMC Psychiatry. 2023 Sep 6;23(1):658. doi: 10.1186/s12888-023-05151-7. PMID 37674135
- [Derived] Axelsson E, Andersson E, Ljotsson B, Bjorkander D, Hedman-Lagerlof M, Hedman-Lagerlof E. Effect of Internet vs Face-to-Face Cognitive Behavior Therapy for Health Anxiety: A Randomized Noninferiority Clinical Trial. JAMA Psychiatry. 2020 Sep 1;77(9):915-924. doi: 10.1001/jamapsychiatry.2020.0940. PMID 32401286
- [Derived] Axelsson E, Lindsater E, Ljotsson B, Andersson E, Hedman-Lagerlof E. The 12-item Self-Report World Health Organization Disability Assessment Schedule (WHODAS) 2.0 Administered Via the Internet to Individuals With Anxiety and Stress Disorders: A Psychometric Investigation Based on Data From Two Clinical Trials. JMIR Ment Health. 2017 Dec 8;4(4):e58. doi: 10.2196/mental.7497. PMID 29222080

DOCUMENTS (1):
  • Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT02314065/SAP_000.pdf